CLINICAL TRIAL: NCT04645251
Title: Polycystic Liver Disease Registry (UK)
Acronym: PLD
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 228220
Record Dates: First submitted 2020-11-11; First posted 2020-11-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Liver Disease
MeSH Terms: conditions — Polycystic liver disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentre, observational registry studying the natural course of polycystic liver disease.

DETAILED DESCRIPTION:
The Polycystic Liver Disease (PLD) registry (UK) is the UK specific part of an international, multicentre, observational registry. The overall international PLD registry is led by Radboud University Medical Center, Nijmegan, Netherlands. Note- please direct any queries about the international registry to the team at Radboud University Medical Center.

All patients with Polycystic Kidney Disease (PKD) with PLD or patients with Isolated (without PKD) Polycystic Liver Disease are eligible for inclusion (>10 liver cysts).

Data will be collected prospectively and retrospectively including a specific validated PLD questionnaire (PLD-Q).

This registry provides us insight in patient characteristics, risk factors, symptoms, quality of life and treatment strategies in the biggest international PLD cohort so far. Results of this registry will be published and shared at national and international congresses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PLD with more than 10 liver cysts
* Patients with PKD and PLD with more than 10 liver cysts

Exclusion Criteria:

* Patients with PKD or PLD with less than 10 liver cysts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mixture of adult patients with PKD and PLD
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Map the natural course of PLD | 10 years
  To establish the demographics, presence and severity of symptoms (quantified using the validated PLD-Q questionnaire), liver cyst characteristics on imaging (assessed using Qian's classification), biochemical marker abnormalities (including gamma-glutamyl transferase and alkaline phosphatase), rate and nature of complications, need for treatment, change in liver volume in patients with PLD. This data will be collected retrospectively and prospectively from clinical records and the PLD-Q questionnaire.

SECONDARY OUTCOMES:
Assess quality of life using the validated PLD questionnaire (PLD-Q) | 10 years
  The PLD-Q questionnaire consists of 18 items assessing symptom frequency and severity. It gives a score (0-100) based on the patient's answers with a higher score indicating more severe, symptomatic disease with a poorer quality of life.
Elucidate risk factors for developing a complication in PLD | 10 years
  For patients that develop a complication of PLD (including jaundice, abdominal hernia, features of portal hypertension, cyst haemorrhage and cyst infection) we will look through their clinical record to establish if there any risk factors which are common to those with a complication (e.g. age, gender, medications, cyst phenotype).
Elucidate elements that affect PLD progression | 10 years
  For patients that have a worsening of their PLD (based on increasing symptoms as per the PLD-Q questionnaire, development of complications or need for treatment) we will look through their clinical records to establish if there any elements which are common to those with progressive disease (e.g. age, gender, medications).
Compare effectiveness of different therapies | 10 years
  For patients who have had or require treatment for PLD we will compare the effectiveness of that treatment based on change in symptoms (based on PLD-Q questionnaire), recurrence of symptoms, development of complications or need for further treatment.
Determine whether rate of liver growth can be used to predict disease progression | 10 years
  Liver growth rate will be determined using change in liver volume on serial radiology imaging. This will be compared against patients symptoms (measured via PLD-Q questionnaire), development of complications and need for treatment to establish whether there is a correlation in rate of liver growth and disease progression

CONTACTS AND LOCATIONS:
Locations (2):
- Radboud University Medical Center, Nijmegen, Netherlands
- Portmouth Hospitals University NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be shared with research team at Radboud University Medical Center, Nijmegen, Netherlands.
Supporting Information: Study Protocol, CSR
Time Frame: Anonymised data will be stored for 15 years

REFERENCES:
- [Background] Neijenhuis MK, Gevers TJ, Hogan MC, Kamath PS, Wijnands TF, van den Ouweland RC, Edwards ME, Sloan JA, Kievit W, Drenth JP. Development and Validation of a Disease-Specific Questionnaire to Assess Patient-Reported Symptoms in Polycystic Liver Disease. Hepatology. 2016 Jul;64(1):151-60. doi: 10.1002/hep.28545. Epub 2016 Apr 15. PMID 26970415
- [Background] van Aerts RMM, van de Laarschot LFM, Banales JM, Drenth JPH. Clinical management of polycystic liver disease. J Hepatol. 2018 Apr;68(4):827-837. doi: 10.1016/j.jhep.2017.11.024. Epub 2017 Nov 24. PMID 29175241
- [Background] Qian Q, Li A, King BF, Kamath PS, Lager DJ, Huston J 3rd, Shub C, Davila S, Somlo S, Torres VE. Clinical profile of autosomal dominant polycystic liver disease. Hepatology. 2003 Jan;37(1):164-71. doi: 10.1053/jhep.2003.50006. PMID 12500201